CLINICAL TRIAL: NCT01151826
Title: Measurement of Physical and Biochemical Markers of Reperfusion Edema During Primary Graft Dysfunction Following Lung Transplantation. Assessment of Their Diagnosis and Prognosis Values
Brief Title: Quantifying Physical and Biochemical Factors That Contribute to Primary Graft Dysfunction After Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, directeur de la Direction de la Recherche Clinique et des Innovations, University Hospital, Strasbourg, France
Other Study IDs: 4714
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Primary Graft Dysfunction
Keywords: Lung transplantation; Primary Graft Dysfunction; Extravascular Lung Water; Receptor for Advanced Glycation Endproducts (RAGE); Intercellular Adhesion Molecule-1 (ICAM-1)
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary graft dysfunction (PGD or lung reperfusion edema) complicates 10 to 20% of lung transplantations and leads to severe early and late postoperative complications. Its pathophysiology remains unclear but may involve graft ischemia-reperfusion, increased vascular permeability, pneumocyte dysfunction and finally alveolar flooding that impair gas exchange and blood oxygenation.Its substrate, namely extravascular lung water (EVLW), can now be clinically measured with minimally invasive Intensive Care Unit monitors (PiCCO2®, Pulsion Medical Systems) that also provides a physical estimate of pulmonary vascular permeability (PVPI). Similarly, biochemical correlates of vascular permeability (ICAM-1) and pneumocyte dysfunction (RAGE) can now be measured in plasma samples. Our study aims at quantifying physical and biochemical markers of PGD and assess their diagnosis and prognosis values.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipient
* Age > 18 years
* Signed informed consent
* Social security affiliation

Exclusion Criteria:

* Age<18
* Pregnancy or lactation
* Contraindication to femoral arterial catheterization
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients cared for in Surgical Intensive Care Unit in Strasbourg University Hospital, France
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and prognosis values of extravascular lung water (EVLW) and pulmonary vascular permeability index (PVPI). | H0 (At started lung transplantation), H6, H12, H24, H48, H72 after lung transplantation

SECONDARY OUTCOMES:
Diagnosis and prognosis values of receptor for advanced glycation endproducts (RAGE) and intercellular adhesion | H0 (At started lung transplantation), H6, H12, H24, H48, H72 after lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Julien Pottecher, MD, Study Director — Service d'Anesthésie-Réanimations chirurgicales - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg Strasbourg, France
Locations (4):
- France (4):
  - Service d'Anesthésie-Réanimations chirurgicales - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Chirurgie thoracique - Nouvel Hôpital Civil - 1, Place de l'hôpital, Strasbourg
  - Service de Physiologie et d'Explorations fonctionnelles - Nouvel Hôpital Civil - 1, Place de l'hôpital, Strasbourg
  - Service de Pneumologie - Nouvel Hôpital Civil -1, Place de l'hôpital, Strasbourg

REFERENCES:
- [Derived] Pottecher J, Roche AC, Degot T, Helms O, Hentz JG, Schmitt JP, Falcoz PE, Santelmo N, Levy F, Collange O, Uring-Lambert B, Bahram S, Schaeffer M, Meyer N, Geny B, Lassalle P, Diemunsch P, Massard G, Kessler R, Steib A; Groupe de Transplantation Pulmonaire des Hopitaux Universitaires de Strasbourg. Increased Extravascular Lung Water and Plasma Biomarkers of Acute Lung Injury Precede Oxygenation Impairment in Primary Graft Dysfunction After Lung Transplantation. Transplantation. 2017 Jan;101(1):112-121. doi: 10.1097/TP.0000000000001434. PMID 27495752